CLINICAL TRIAL: NCT06910124
Title: Alpe d'Huez Study: A Parallel Two-Cohort Study of Linvoseltamab in Addition to Lenalidomide (L2) During Maintenance Therapy of NDMM to Deepen Responses or Redrive MRD Negativity After Relapse
Brief Title: Linvoseltamab in Addition to Lenalidomide (L2) During Maintenance Therapy of NDMM to Deepen Responses or Redrive MRD Negativity After Relapse
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dickran Kazandjian, MD (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Dickran Kazandjian, MD, Professor of Clinical, University of Miami
Organization: University of Miami (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20241138
Record Dates: First submitted 2025-03-27; First posted 2025-04-04 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma
Keywords: Newly Diagnosed Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 - Linvoseltamab Treatment Group (Experimental): Participants in this group are currently receiving lenalidomide maintenance therapy for ≤12 months will have linvoseltamab added to the lenalidomide maintenance therapy and receive treatment with the combination for up to 24 cycles.
  Total participation duration is up to 4.5 years
  Interventions: Biological: Linvoseltamab; Drug: Lenalidomide
- Cohort 2 - Lenalidomide Treatment Group (Experimental): Participants in this group are currently receiving lenalidomide maintenance therapy but have relapsed disease within 12 months of starting maintenance will have Linvoseltamab added to lenalidomide maintenance and receive treatment with the combination for up to 24 cycles.
  Total participation duration is up to 4.5 years
  Interventions: Biological: Linvoseltamab; Drug: Lenalidomide

INTERVENTIONS:
Biological: Linvoseltamab — Participants will receive Linvoseltamab intravenously (IV) according to the following schedule and regimen, for up to 24 cycles, each cycle lasting 28 days:
  * Cycle 1 Day 1: 5mg
  * Cycle 1 Day 8: 25mg
  * Cycle 1 Days 15, 22: 100mg
  * Cycles 2 and 3, Days 1, 8, 15, 22: 100mg
  * Cycles 3 and 6, Days 1 and 15: 100mg
  * Cycles 7 through 24: 100mg
Drug: Lenalidomide — Participants will take 10mg of Lenalidomide maintenance therapy standard of care by mouth daily from days 1 through 21 of each 28 day cycle of Linvoseltamab therapy. Lenalidomide therapy will begin on Cycle 2 Day 1 of Linvoseltamab therapy.

SUMMARY:
The purpose of this study is to determine whether giving linvoseltamab with lenalidomide during maintenance treatment to participants with multiple myeloma will:

1. Get rid of any residual multiple myeloma cells in participants' bodies which is known as minimal residual disease negative (MRD-) status. For participants that start the study with residual multiple myeloma cells in participants' bodies: to determine how long you remain MRD-.
2. Increase the length of time that participants' disease is controlled. For participants with relapsed disease, to determine whether participants can re-attain MRD- status.
3. Increase the length of time that participants' disease responds to treatment.

The researchers also want to find out the effects that linvoseltamab has on participants and participants' condition.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of newly-diagnosed multiple myeloma (NDMM) per International Myeloma Working Group (IMWG) documented initially prior to any treatment (Kumar et al., 2016).
2. Documentation of having received a triplet or quadruplet based initial combination therapy containing at least two of the following: Immunomodulatory drug (IMiD), proteosome inhibitor (PI), and/or anti-cluster of differentiation 38 (anti-CD38).
3. Documentation of receiving induction therapy with or without high-dose melphalan with autologous stem cell transplant (HDM-ASCT) and receiving lenalidomide maintenance therapy ≤ 12 months.

   1. Cohort 1: at the time of assessment, the patient's current response is a partial response (PR), very good partial response (VGPR), or complete response (CR) but MRD+ by the FDA-cleared next-generation sequencing (NGS) Adaptive clonoseq assay.
   2. Cohort 2: at the time of assessment, the patient has a relapse from their initial complete response (CR) (<CR response are ineligible) post induction but do not meet criteria for IMWG progression (eg, patients who no longer meet criteria for CR but whose M-protein is ≤ 0.5 g/dL and/or immunofixation has turned positive, and/or have converted to MRD+ by the FDA-cleared NGS Adaptive clonoseq assay).
4. Eastern Cooperative Oncology Group Performance Status (ECOG PS) ≤ 3 (Appendix A)
5. Adequate organ function

   1. Absolute neutrophil count (ANC) ≥ 1000/microlitre (unless patient has ethnic neutropenia)
   2. Platelets ≥ 50,000/microlitre
   3. Hemoglobin ≥ 8 g/dL (transfusions permitted)
   4. Serum total bilirubin ≤ 1.5 X upper limit of normal (ULN) or direct bilirubin ≤ ULN for patients with total bilirubin levels > 1.5 ULN (except patients with Gilbert's syndrome who must have a total bilirubin of < 3 X ULN)
   5. Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase (SGOT)) and alanine aminotransferase (ALT) (serum glutamic-pyruvic transaminase (SGPT)) ≤ 3 X ULN
   6. Serum creatinine ≤ 1.5 X ULN (except if due to myeloma) or calculated estimated glomerular filtration rate (eGFR)/creatinine clearance (CrCl) (by Chronic Kidney Disease Epidemiology Collaboration, Modification of Diet in Renal Disease, or Cockcroft-Gault) ≥ 15 mL/min/1.73 m2
6. Female patients of childbearing potential must have a negative serum pregnancy test at Screening. Female patients of childbearing potential and fertile male patients who are sexually active with a female of childbearing potential must use highly effective methods of contraception throughout the study and for 90 days following the last dose of study treatment.
7. Willing and able to provide written informed consent in accordance with federal, local, and institutional guidelines. The patient must provide informed consent prior to the first screening procedure.
8. Willing and able to comply with clinic visits and study-related procedures.

Exclusion Criteria:

1. Patients who have received prior systemic therapies for Multiple Myeloma (MM) other than initial IMiD/PI/anti CD38/HDM-ASCT-based combination therapy.

   * Treatment with corticosteroids for MM or other indications is permitted.
   * Prior radiation therapy and surgery is permitted.
2. Patients who are receiving any other investigational agents unless deemed not to interfere with the study by the Principal Investigator (PI).
3. Patients who receive a live attenuated vaccine within 4 weeks of scheduled study treatment administration.
4. Contraindication to any concomitant medication, including those medications administered for infusion reaction, antiviral, antibacterial, anticoagulation, tumor lysis, or hydration prophylaxis given prior to therapy.
5. Patient has any of the following:

   * a. Human immunodeficiency virus (HIV)-positive with 1 or more of the following: i. History of acquired immune deficiency syndrome (AIDS)-defining conditions Cluster of differentiation 4 count < 350 cells/mm3 ii. Detectable viral load during screening or within 6 months prior to screening iii. Not receiving highly active anti-retroviral therapy iv. Had a change in antiretroviral therapy within 6 months of the start of screening v. Receiving antiretroviral therapy that may interfere with study treatment as assessed after discussion with the PI
   * b. Hepatitis B infection (ie, hepatitis B surface antigen (HBsAg) or hepatitis B virus (HBV) DNA positive). Patients with resolved infection (ie, patients who are HBsAg negative but positive for antibodies to hepatitis B core antigen [anti-Hepatitis-C] and/or antibodies to hepatitis B surface antigen [anti-HBs]) must be screened using real-time polymerase chain reaction (PCR) measurement of HBV deoxyribonucleic acid (DNA) levels. Those who are PCR positive will be excluded. In the event the infection status is unclear, quantitative viral levels are necessary to determine the infection status. Exception: Patients with serologic findings suggestive of HBV vaccination (anti HBs positivity as the only serologic marker) AND a known history of prior HBV vaccination do not need to be tested for HBV DNA by PCR.

     c. Active hepatitis C (HCV) infection as measured by positive HCV-ribonucleic acid (RNA) testing. Participants with a history of HCV antibody positivity must undergo HCV-RNA testing. If a participant with history of chronic hepatitis C infection (defined as both HCV antibody and HCV RNA positive) completed antiviral therapy and has undetectable HCV RNA 12 weeks following the completion of therapy, the participant is eligible for the study.
6. History of allergic reactions attributed to compounds of similar chemical or biologic composition to the experimental agents used in study.
7. Female patient refuses to discontinue breastfeeding her infant during study treatment or within 3 months after receiving the last dose of study treatment.
8. Participant plans to father a child while enrolled in this study or within 3 months after the last dose of study treatment.
9. Presence of the following cardiac conditions:

   1. New York Heart Association stage III or IV congestive heart failure
   2. Myocardial infarction or coronary artery bypass graft ≤ 3 months prior to study enrollment
   3. History of clinically significant ventricular arrhythmia or unexplained syncope, not believed to be vasovagal in nature or due to dehydration Uncontrolled cardiac arrhythmia or clinically significant electrocardiogram (ECG) abnormalities
   4. Unstable or uncontrolled disease/condition related to or affecting cardiac function (eg, unstable angina)
10. Uncontrolled intercurrent illness including but not limited to ongoing or active infection, venous thromboembolic disease, hemorrhage, pulmonary fibrosis, pneumonitis, active autoimmune disease or a documented history of autoimmune disease with the exception of vitiligo, type I diabetes, and prior autoimmune thyroiditis that is currently euthyroid based on clinical symptoms and laboratory testing, or psychiatric illness/social situations within 2 weeks that would limit compliance with study requirements.
11. History of neurodegenerative condition, central nervous system (CNS) movement disorder, or patients with a history of seizure within 12 months prior to study enrollment are excluded unless deemed clinically not significant risk by the PI.
12. Active malignancy other than MM requiring treatment in the past 6 months. Malignancies treated within the past 6 months that are considered cured with minimal risk of recurrence are allowed.
13. Have any condition that, in the opinion of the Investigator, would compromise the well-being of the patient or the study or prevent the patient from meeting or performing study requirements.
14. Patients with impaired decision-making capacity will not be enrolled on this trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-12-02 (Actual); Primary Completion 2032-12-02 (Estimated); Study Completion 2032-12-02 (Estimated)

PRIMARY OUTCOMES:
Minimum Residual Disease Negative Conversion Rate | 12 months
  The number of patients who experience MRD negativity (10^-5 sensitivity by 12 cycles of linvoseltamab (MRD conversion rate) will be determined by dividing this number of MRD negative responses by the total number of evaluable patients.
  MRD negativity rate (<10^-5) by 12 cycles of linvoseltamab

SECONDARY OUTCOMES:
Minimum Residual Disease Negative Conversion Rate | 6 months
  The number of patients who experience MRD negativity (10^-5 sensitivity) by 6 months of Linvoseltamab (MRD conversion rate) will be determined by dividing this number of MRD negative responses by the total number of evaluable patients.
Sustained MRD Negativity Rate | Up to 2 years
  The sustained rate of MRD-negativity, at a sensitivity of <10^-5, among participants will be reported. The duration of time in months measured from the first time the participant achieves an MRD-negative bone marrow (BM) biopsy result until the time the participant has relapsed from MRD-negativity objectively documented with an MRD-positive BM result.
Overall Response Rate | Up to 12 months
  The number of participants achieving stringent complete response (sCR), complete response (CR), very good partial response (VGPR), partial response or minimal response (MR) to study therapy. Multiple myeloma (MM) response assessments will be made in accordance with modified International Myeloma Working Group (IMWG) 2016 response criteria.
Best Overall Response (BOR) | Up to 12 months
  The best overall response is defined as the best response by the percentage of participants recorded from start of study therapy until the completion of 12 cycles of study therapy. Multiple myeloma (MM) response assessments will be made in accordance with modified International Myeloma Working Group (IMWG) 2016 response criteria.
Duration of Response (DOR) | Up to 4.5 years
  Duration of response is defined as the elapsed time in months from the time the criteria are met for achieving partial response (PR) or better until the time of progressive disease (PD) is objectively documented. Multiple myeloma (MM) response assessments will be made in accordance with modified International Myeloma Working Group (IMWG) 2016 response criteria.
Progression-Free Survival (PFS) | Up to 4.5 years
  PFS is defined as the elapsed time in months from the start of study therapy until first documented progressive disease (PD). Multiple myeloma (MM) response assessments will be made in accordance with modified International Myeloma Working Group (IMWG) 2016 response criteria.
Overall Survival (OS) | Up to 4.5 years
  Overall survival (OS) is defined as the elapsed time in months from start of study therapy to death or censoring at last known time point that participant was known to be alive (may be based on clinic visit or phone call, etc.)
Number of Participants Experiencing Treatment-related Adverse Events | Up to 27 months
  The number of participants experiencing all Grade and Grade ≥3 treatment-related adverse events will be recorded. Adverse events will be assessed using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0, per physician discretion.

CONTACTS AND LOCATIONS:
Overall Officials: Dickran Kazandjian, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No